CLINICAL TRIAL: NCT02631837
Title: Hysterectomy for Benign Gynaecological Disease by Natural Orifice Transluminal Endoscopic Surgery or Laparoscopy
Brief Title: Hysterectomy by Transabdominal Laparoscopy or NOTES
Acronym: HALON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imelda Hospital, Bonheiden (Other)
Responsible Party: Principal Investigator, Dr Jan Baekelandt, MD, Dr, Imelda Hospital, Bonheiden
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B689201526261
Record Dates: First submitted 2015-12-09; First posted 2015-12-16 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Uterine Diseases
Keywords: NOTES; Laparoscopic surgery
MeSH Terms: conditions — Uterine Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vNOTES hysterectomy (Experimental): vaginal Natural Orifice Transluminal Endoscopic Surgery
  Interventions: Procedure: vNOTES hysterectomy
- LSC hysterectomy (Active Comparator): Laparoscopic hysterectomy
  Interventions: Procedure: LSC hysterectomy

INTERVENTIONS:
Procedure: vNOTES hysterectomy — Surgical removal of the uterus by Natural Orifice Transluminal Endoscopic Surgery using a colpotomy
  Arms: vNOTES hysterectomy
Procedure: LSC hysterectomy — Surgical removal of the uterus by transabdominal laparoscopy
  Arms: LSC hysterectomy

SUMMARY:
Objective: To randomly compare hysterectomy by vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) versus laparoscopy uterus in women with benign gynecological pathology.

Study design: Randomized controlled/single center/single-blinded/parallel-group/non-inferiority/efficacy trial.

Study population: All women aged 18 to 70 years regardless of parity with a non-prolapsed uterus and a benign indication for hysterectomy.

Primary study outcome parameters: successful removal of the uterus by the intended technique.

Secondary outcomes: the proportion of women admitted to the in-hospital ward; postoperative pain scores; the total amount of analgesics used; postoperative infection; per- or postoperative complications; hospital readmission rates; duration of the surgical procedure; incidence and intensity of dyspareunia; sexual wellbeing; health-related quality of life; costs.

DETAILED DESCRIPTION:
l1.Objectives of the HALON Trial The primary research questions of this IDEAL stage 2b efficacy trial are as follows: is a vNOTES (vaginal Natural Orifice Transluminal Endoscopic Surgery) hysterectomy at least as effective compared to the standard transabdominal laparoscopic approach (LSC) for removing a non-prolapsed uterus without the need for conversion to an alternative approach? (non inferiority design)

Secondary research questions are:

* Do more women treated by vNOTES prefer to leave the day care unit on the day of surgery compared to LSC?
* Do women treated by vNOTES suffer from less pain compared to women treated by LSC in the first postoperative week?
* Is the removal of a uterus by vNOTES faster compared to LSC?
* Does a vNOTES cause more pelvic infection or other complications compared to LSC?
* Does a vNOTES result in more hospital readmissions within 6 weeks after surgery compared to LSC?
* Does a vNOTES approach result in more women reporting dyspareunia, less sexual wellbeing or less health-related quality of life at 3 or 6 months after surgery when compared to women treated by LSC?
* What are the direct and indirect costs up to 6 weeks after the surgical intervention of a vNOTES compared to LSC? 2. TRIAL DESIGN 2.1. Design A single center, single-blinded, parallel group randomized, non-inferiority efficacy trial.

2.2. Simple pilot randomized trial. 2.3. Time schedule Based upon the mean number of hysterectomies performed annually for benign gynecological disease at the department of Obstetrics and Gynecology of the participating center (168) the investigators estimate that the duration of recruitment will be 12 months. Based upon the follow up (6 months) and the period of analysis/reporting (3 months) the total study period will be 2 years.

2.4. Participating center Department of Obstetrics and Gynecology Imeldahospital Imeldalaan 9 2820 Bonheiden Belgium 3. ELIGIBILITY, CONSENT AND RANDOMIZATION 3.1. Screening and consent prior to surgery All women aged 18 to 70 years, regardless of parity, with a non-prolapsed uterus in need of a hysterectomy for benign indication are eligible for inclusion.

3.2. Determining eligibility All women aged 18 to 70 years, regardless of parity, with a non-prolapsed uterus in need of a hysterectomy for benign indication who provide consent to participation are eligible in the HALON trial and will be randomized before the procedure.

3.3. Randomization If the woman is eligible for the HALON trial, the trial secretary will obtain a randomized allocation the day before surgery. This will be done using a randomization list generated by a free computer software program offered by Research Randomizer (https://www.randomizer.org). The random sequence generation will be concealed using sequentially numbered opaque sealed envelopes. The envelope will be opened by the nurse assistant the day before surgery for practical logistic reasons.

3.4. Patients with strong preference for treatment A minority of women will express a clear preference for one of both treatments (e.g. strong desire to have no scar) and for this reason will not wish to be randomized between surgical treatments. To investigate how outcomes vary by choice, these women could be followed up in exactly the same way as for those women randomized into the HALON trial. A formal non-randomized follow-up of these women will not be done for logistical reasons.

3.5. Stratification of randomization A blocked randomization procedure will be used to avoid chance imbalances for the parameter 'uterine size'.

4. TREATMENT ALLOCATIONS 4.1. Surgical procedures The principal investigator, who has training and experience in both laparoscopy and NOTES, will perform all surgical procedures. He is therefore not blinded. All vNOTES participants will be blinded by three superficial non-therapeutic or "mock" skin incisions similar to those done with the laparoscopic technique.

4.1.1 vNOTES hysterectomy This is the surgical procedure done in the intervention arm of the HALON trial. 4.1.2 LSC hysterectomy This is the surgical procedure done in the control arm of the HALON trial. 5. FOLLOW-UP AND OUTCOME MEASURES 5.1. Clinical assessments 5.1.1 Format PROMs (Patient reported outcomes) will be collected using a postal questionnaire, which will include a combination of disease specific (Pain on sexual intercourse measured by VAS scale and SSFS Scale) and generic measurement instruments (EQ-5D).

The postal questionnaires will be sent from the HALON Trial Office with postage paid envelopes two weeks before the due date. Reminders will be sent to patients if the questionnaire is not returned within one week of the due date and attempts will be made to contact the patient by phone if the questionnaire is not returned by two weeks after the due date.

5.1.2 Timing of assessments The primary outcome will be measured clinically at the end of the surgical procedure. In addition PROMs will take place at baseline (pain on sexual intercourse, health-related quality of life and sexual well being), the evening of the surgical intervention (in-hospital admission), during the first postoperative week (pain by VAS scores and analgetic drugs) and at 3 and 6 months (dyspareunia/ sexual well being/health related quality of life). Clinical physician assessment will take place the evening of the surgical intervention (in-hospital admission) and during the first six weeks following surgery (pelvic infection, surgical complications, hospital readmission rate).

5.2. Primary clinical outcome measure The proportion of women successfully treated by removing the uterus by the intended approach without conversion to another approach, using a dichotomous outcome measure, will be used as a measure of efficacy.

5.3. Secondary clinical outcome measures

The following secondary outcomes will be measured:

* The proportion of women addmitted in-hospital for at least one night observation based on their own preference, as a dichotomous outcome.
* Postoperative pain scores, as an ordinal outcome, measured using a Visual Analogue Scale (VAS) twice daily from day 1 till 7 self-reported by the participating women. The VAS scores range from 0= no pain to 10= worst imaginable pain.
* Postoperative pain defined by the total amount of analgesics used as described in the standardized pain treatment protocol, as a continuous outcome.
* Postoperative infection as a dichotomous outcome.
* Per- or postoperative complications according to the Clavien- Dindo classification detected during the first six weeks of surgery, as a dichotomous outcome.
* The number of women readmitted to hospital within 6 weeks following surgery.
* Incidence and intensity of dyspareunia recorded by the participants at baseline, 3 and 6 months by self-reporting using a simple questionnaire and a Visual Analogue Scale (VAS) scale, as a dichotomous and ordinal outcome. The VAS scores range from 0= no pain to 10= worst imaginable pain.
* Sexual wellbeing at baseline, at 3 and 6 months by self-reporting the Short Sexual Functioning Scale (SSFS). The SSFS is a questionnaire with 7 multiple choice open ended questions.
* Health related quality of life, at baseline, at 3 and 6 months by self-reporting the EQ-5D-3L scale. The EQ-5D-3L scale is a questionnaire on 5 domains with 3 open ended questions and a scale from 0= worst possible health-related quality of life to 100= best possible health-related quality of life.
* Duration of surgery measured as the time in minutes from the insertion of the bladder catheter to the end of vaginal/abdominal wound closure, as a continuous outcome. 5.4.The direct and indirect costs up to 6 weeks after the hysterectomy of the vNOTES technique compared to LSC.

  6. ACCRUAL AND ANALYSIS 6.1. Sample size The sample size for the primary outcome of this trial has been chosen to give good statistical power to preclude any clinically important inferiority of vNOTES compared to laparoscopy and is based on evidence retrieved from a Dutch prospective cohort study. Based on the power calculations for the primary outcome and assuming a loss-to-follow-up rate of 15% we decided to include 66 study participants in the HALON trial.

6.2. Projected accrual and attrition rates Based upon the mean number of hysterectomies performed annually at the department of Obstetrics and Gynecology of the participating center (168) the investigators anticipate that the duration of recruitment will be 12 months. Based upon the follow up (6 months) and the period of analysis/reporting (3 months) the total study period will be 2 years. First publication will be possible within four years of trial commencement.

The sample size calculations have allowed for a 15% loss to follow up rate. In order to minimize rates of attrition a dedicated research secretary will be employed to optimize recruitment and follow up.

ELIGIBILITY:
Inclusion Criteria:

* All women aged 18 to 70 years regardless of parity, with a non-prolapsed uterus in need of a hysterectomy for benign indication
* Written informed consent obtained prior to surgery

Exclusion Criteria:

* History of rectal surgery
* Suspected rectovaginal endometriosis
* Suspected malignancy
* History of pelvic inflammatory disease, especially prior tubo-ovarian or pouch of Douglas abscess
* Active lower genital tract infection e.g. Chlamydia, N. gonorrhoeae
* Virgo
* Pregnancy
* Failure to provide written informed consent prior to surgery

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Baekelandt, MD, Principal Investigator — Imelda Hospital, Bonheiden
Locations (1):
- Imelda Hospital, Bonheiden, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No
Interim analyses of major endpoints will be supplied, in strict confidence, to an independent Data Monitoring and Ethics Committee (DMEC) along with updates on results of other related studies, and any other analyses that the DMEC may request.

REFERENCES:
- [Background] Reynders A, Baekelandt J. Adnexectomy by Poor Man's Transvaginal NOTES. Gynecol Surg 2015; 12: 207-11
- [Background] Van Peer S, Baekelandt J. Natural orifice transluminal endoscopic surgery (NOTES) salpingectomy for ectopic pregnancy: a first series demonstrating how a new surgical technique can be applied in a low-resource setting. Gynecol Surg 2015; 12: 299-302
- [Background] Baekelandt J, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol BW, Bosteels JJ. HALON-hysterectomy by transabdominal laparoscopy or natural orifice transluminal endoscopic surgery: a randomised controlled trial (study protocol). BMJ Open. 2016 Aug 12;6(8):e011546. doi: 10.1136/bmjopen-2016-011546. PMID 27519922
- [Background] Baekelandt JF, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol B, Bosteels J. Hysterectomy by transvaginal natural orifice transluminal endoscopic surgery versus laparoscopy as a day-care procedure: a randomised controlled trial. BJOG. 2019 Jan;126(1):105-113. doi: 10.1111/1471-0528.15504. PMID 30325565
- [Result] Su H, Yen CF, Wu KY, Han CM, Lee CL. Hysterectomy via transvaginal natural orifice transluminal endoscopic surgery (NOTES): feasibility of an innovative approach. Taiwan J Obstet Gynecol. 2012 Jun;51(2):217-21. doi: 10.1016/j.tjog.2012.04.009. PMID 22795097
- [Result] Lee CL, Wu KY, Su H, Wu PJ, Han CM, Yen CF. Hysterectomy by transvaginal natural orifice transluminal endoscopic surgery (NOTES): a series of 137 patients. J Minim Invasive Gynecol. 2014 Sep-Oct;21(5):818-24. doi: 10.1016/j.jmig.2014.03.011. Epub 2014 Mar 25. PMID 24681063
- [Result] Atallah S, Martin-Perez B, Albert M, Schoonyoung H, Quinteros F, Hunter L, Larach S. Vaginal Access Minimally Invasive Surgery (VAMIS): A New Approach to Hysterectomy. Surg Innov. 2015 Aug;22(4):344-7. doi: 10.1177/1553350614560273. Epub 2014 Nov 27. PMID 25432882
- [Result] Yang YS, Kim SY, Hur MH, Oh KY. Natural orifice transluminal endoscopic surgery-assisted versus single-port laparoscopic-assisted vaginal hysterectomy: a case-matched study. J Minim Invasive Gynecol. 2014 Jul-Aug;21(4):624-31. doi: 10.1016/j.jmig.2014.01.005. Epub 2014 Jan 21. PMID 24462594
- [Result] Wang CJ, Huang HY, Huang CY, Su H. Hysterectomy via transvaginal natural orifice transluminal endoscopic surgery for nonprolapsed uteri. Surg Endosc. 2015 Jan;29(1):100-7. doi: 10.1007/s00464-014-3639-y. Epub 2014 Oct 1. PMID 25270610
- [Result] Baekelandt J. Total Vaginal NOTES Hysterectomy: A New Approach to Hysterectomy. J Minim Invasive Gynecol. 2015 Sep-Oct;22(6):1088-94. doi: 10.1016/j.jmig.2015.05.015. Epub 2015 May 22. PMID 26009278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 9, 2015, and February 23, 2017, 194 women were screened for eligibility
Period: Overall Study
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants included were women.
Groups:
- Total: Total of all reporting groups
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Full Range); unit: Years] — Age of the participants in years
  Years | 46 [24 to 65] | 49 [34 to 68] | 47 [24 to 68]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 35 | 35 | 70
Body Mass Index [Mean (Full Range); unit: kg/m²] | 26.6 [17.7 to 44.1] | 26.4 [18.6 to 42.9] | 26.5 [17.7 to 44.1]
Number of vaginal births [Mean (Full Range); unit: number of vaginal births] | 1.4 [0 to 4] | 1.3 [0 to 3] | 1.4 [0 to 4]
Prior abdominal surgery [Count of Participants; unit: Participants] | 20 | 16 | 36
Prior Caesarean section [Count of Participants; unit: Participants] | 8 | 5 | 13
Uterine weight [Mean (Full Range); unit: grams] | 206.2 [44.0 to 788.0] | 177.3 [28.0 to 590.0] | 191.7 [28.0 to 788.0]
Pain vagina sexual intercourse [Count of Participants; unit: Participants] | 15 | 6 | 21
Pain abdomen sexual intercourse [Count of Participants; unit: Participants] | 12 | 8 | 20
Health-related quality of life [Mean (Full Range); unit: units on a scale] — The reported values for the health-related quality of life are self-reported values using the VAS part of the two part EuroQoL EQ-5D-3L questionnaire. The scale ranges from 0 (worst quality) to 100 (best quality).
  units on a scale | 74.6 [20 to 100] | 76.8 [20 to 100] | 75.7 [20 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Successful Removal of the Uterus Without Conversion to Another Technique
Description: Successful removal of the uterus without conversion to another technique with or without morcellation
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
Participants | 35 | 35
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Non-Inferiority — Our hypothesis was that women would accept a higher conversion rate of 15% for vNOTESbased on a telephone interview of 10 women treated by total vaginal NOTES hysterectomy. Women were asked to choose among ﬁve cut-off rates (5, 10, 15, 20 or 25%). Most women indicated 15%. We would conclude non-inferiority when the upper limit of the one-sided 95% conﬁdence interval for the difference in the proportions of women between both comparisons would be below 15%; p = 0.0221, Farrington-Manning — The Farrington-Manning test for non-inferiority was performed with 5% significance level and yielded P = 0.0221 in a sensitivity analysis assuming one conversion in the vNOTES and 0 conversions in the laparoscopy group

2. Secondary Outcome: Admission in Hospital for at Least One Night Observation
Description: The number of women admitted in-hospital for at least one night observation based on their own preference after discharge from the day care unit, as a dichotomous outcome. The decision to discharge or to admit to hospital for the night will be based solely on the choice of the woman to return home the same day or stay overnight.
Time Frame: Measured on the day of the surgical intervention
Measure: Count of Participants; unit: Participants
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
Participants | 8 | 20
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p = 0.007, Fisher Exact; Risk Difference (RD) = -0.34, 95% CI 2-sided [-0.56 to -0.13]
Statistical Analysis 2: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p = 0.007, Fisher Exact

3. Secondary Outcome: Postoperative Pain Scores
Description: Postoperative pain scores, as an ordinal outcome, measured using a Visual Analogue Scale (VAS) twice daily (morning and evening) from day 1 till 7 selfreported by the participating women. VAS scores from 0 to 10 with 0 = no pain and 10= worst pain ever imaginable.
Time Frame: The first seven days after the surgical intervention
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
units on a scale
  mean pain VAS score day 1 morning | 3.629 [2.877 to 4.380] | 4.200 [3.449 to 4.951]
  mean pain VAS score day 1 evening | 3.486 [2.815 to 4.157] | 4.456 [3.783 to 5.129]
  mean pain VAS score day 2 morning | 2.486 [1.876 to 3.096] | 3.543 [2.933 to 4.153]
  mean pain VAS score day 2 evening | 2.514 [1.947 to 3.082] | 3.343 [2.775 to 3.910]
  mean pain VAS score day 3 morning | 1.800 [1.261 to 2.339] | 2.800 [2.261 to 3.339]
  mean pain VAS score day 3 evening | 1.857 [1.335 to 2.379] | 2.914 [2.392 to 3.436]
  mean pain VAS score day 4 morning | 1.257 [0.746 to 1.769] | 2.286 [1.774 to 2.797]
  mean pain VAS score day 4 evening | 1.371 [0.867 to 1.876] | 2.457 [1.952 to 2.962]
  mean pain VAS score day 5 morning | 1.143 [0.643 to 1.642] | 1.914 [1.415 to 2.414]
  mean pain VAS score day 5 evening | 1.057 [0.562 to 1.553] | 2.086 [1.590 to 2.581]
  mean pain VAS score day 6 morning | 0.914 [0.421 to 1.407] | 1.914 [1.421 to 2.407]
  mean pain VAS score day 6 evening | 1.086 [0.591 to 1.580] | 2.000 [1.505 to 2.495]
  mean pain VAS score day 7 morning | 1.029 [0.525 to 1.532] | 1.567 [1.060 to 2.074]
  mean pain VAS score day 7 evening | 0.819 [0.290 to 1.348] | 1.693 [1.153 to 2.233]

4. Secondary Outcome: The Use of Analgetic Drugs for Postoperative Pain
Description: Postoperative pain defined by the total amount of analgesics used as described in the standardized pain treatment protocol, as a continuous outcome.
Time Frame: The first week after the surgical intervention
Measure: Mean (Full Range); unit: number of tablets
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
number of tablets | 8.0 [0 to 28] | 13.9 [0 to 50]
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p = 0.006, Mann-Whitney U test; Two-sided test; Mean Difference (Final Values) = -5.9, 95% CI 2-sided [-10 to -1.8]

5. Secondary Outcome: Postoperative Infection
Description: Postoperative infection defined by lower abdominal pain with fever > 38°C and positive clinical signs or laboratory findings, detected during the first six weeks of surgery, as a dichotomous outcome.
Time Frame: The first six weeks after the surgical intervention
Measure: Count of Participants; unit: Participants
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
Participants | 1 | 2
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p = 1.00, Fisher Exact

6. Secondary Outcome: Intra- Operative Complications
Description: Intra- operative complications according to the Clavien- Dindo classification detected during the first six weeks of surgery, as a dichotomous outcome
Time Frame: At the time of the surgical intervention
Measure: Count of Participants; unit: Participants
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
Participants | 1 | 0
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p > 0.05, Fisher Exact

7. Secondary Outcome: Postoperative Complications
Description: Postoperative complications detected during the first six weeks of surgery, as a dichotomous outcome
Time Frame: The first six weeks after the surgical intervention
Measure: Count of Participants; unit: Participants
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
Participants | 3 | 13
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p = 0.009, Fisher Exact; Risk Difference (RD) = -0.29, 95% CI 2-sided [-0.47 to -0.10]

8. Secondary Outcome: Hospital Readmission
Description: The number of women readmitted to hospital within six weeks following surgery, as a dichotomous outcome.
Time Frame: The first six weeks after the surgical intervention
Measure: Count of Participants; unit: Participants
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
Participants | 1 | 6
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p = 0.106, Fisher Exact

9. Secondary Outcome: Duration of the Surgical Intervention
Description: Duration of surgery measured as the time in minutes from the insertion of the bladder catheter to the end of vaginal/ abdominal wound closure, as a continuous outcome
Time Frame: Intraoperative
Measure: Mean (Full Range); unit: minutes
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
minutes | 41.1 [21.0 to 130.0] | 75.1 [40.0 to 189.0]
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p < 0.01, Mann-Whitney U test; Median Difference (Final Values) = -34, 95% CI 2-sided [-46 to -22]

10. Secondary Outcome: Vaginal Pain During Sexual Intercourse at Three Months
Description: Incidence of vaginal dyspareunia recorded by the participants at 3 months by self-reporting using a simple questionnaire.
Time Frame: At 3 months after the surgical intervention
Measure: Count of Participants; unit: Participants
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
Participants | 8 | 9
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p = 0.7604, Arm by time interaction — We tested a treatment arm by time interaction to study changes in differences for the outcomes during the follow-up period. In absence of such an interaction (p>0.05 for the interaction term), the main effect of treatment was tested

11. Secondary Outcome: Vaginal Pain During Sexual Intercourse at Six Months
Description: Incidence of vaginal dyspareunia recorded by the participants at 6 months by self-reporting using a simple questionnaire
Time Frame: At 6 months after the surgical intervention
Measure: Count of Participants; unit: Participants
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
Participants | 5 | 8
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p = 0.3071, Arm by time interaction — [p-value comment as in outcome 10, analysis 1]

12. Secondary Outcome: Pelvic Pain During Sexual Intercourse at Three Months
Description: Incidence of pelvic dyspareunia recorded by the participants at 3 months by self-reporting using a simple questionnaire.
Time Frame: At 3 months after the surgical intervention
Measure: Count of Participants; unit: Participants
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
Participants | 6 | 8
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p = 0.4541, Arm by time interaction — [p-value comment as in outcome 10, analysis 1]

13. Secondary Outcome: Pelvic Pain During Sexual Intercourse at Six Months
Description: Incidence of pelvic dyspareunia recorded by the participants at 6 months by self-reporting using a simple questionnaire.
Time Frame: At 6 months after the surgical intervention
Measure: Count of Participants; unit: Participants
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
Participants | 4 | 5
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p = 0.4514, Arm by time interaction — [p-value comment as in outcome 10, analysis 1]

14. Secondary Outcome: Health-related Quality of Life at Three Months
Description: Health-related quality of life at 3 months by self-reporting the EQ-5D scale.The reported values for the health-related quality of life are self-reported values using the VAS part of the two part EQ-5D-3L questionnaire. The scale ranges from 0 (worst quality) to 100 (best quality).
Time Frame: At 3 months after the surgical intervention
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
score on a scale | 83.8 [40.0 to 100.0] | 79.6 [20.0 to 100.0]
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p = 0.3473, Arm by time interaction — [p-value comment as in outcome 10, analysis 1]

15. Secondary Outcome: Health-related Quality of Life at Six Months
Description: Health-related quality of life at 6 months by self-reporting the EQ-5D scale. The reported values for the health-related quality of life are self-reported values using the VAS part of the two part EQ-5D-3L questionnaire. The scale ranges from 0 (worst quality) to 100 (best quality).
Time Frame: At 6 months after the surgical intervention
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
score on a scale | 87.8 [60.0 to 100.0] | 86.6 [65.0 to 100.0]
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority — We tested a treatment arm by time interaction to study changes in differences for the outcomes during the follow-up period. In absence of such an interaction (p>0.05 for the interaction term), the main effect of treatment was tested; p = 0.3473, Arm by time interaction — [p-value comment as in outcome 10, analysis 1]

16. Secondary Outcome: Sexual Well Being
Description: Sexual wellbeing at baseline, at 3 and 6 months by self-reporting using the SSFS (Short Sexual Function Scale). The SSFS is a questionnaire of 7 open ended questions on sexual wellbeing.
Time Frame: At baseline, 3 months and 6 months after the surgical intervention
Reporting Status: Not Posted, anticipated posting 2024-12

17. Secondary Outcome: Direct Costs
Description: Calculating the comparative direct costs in USD of both techniques up to 6 weeks after the surgical intervention
Time Frame: Up to 6 weeks postoperative
Measure: Mean (Full Range); unit: USD
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
Number analyzed (Participants) | 35 | 35
USD | 3452.2 [2404.6 to 4897.1] | 3933.6 [2120.6 to 6776.2]
Statistical Analysis 1: Comparison: vNOTES Hysterectomy vs LSC Hysterectomy; Test type: Superiority; p = 0.110, Mann-Whitney U test; Mean Difference (Final Values) = -555.8, 95% CI 2-sided [-1,044 to 36]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Intra- or postoperative complications
Arm/Group | vNOTES Hysterectomy | LSC Hysterectomy
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 2/35
Other Adverse Events (participants affected / at risk) | 3/35 | 11/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | vNOTES Hysterectomy (N=35) | LSC Hysterectomy (N=35)
vesicovaginal fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | vNOTES Hysterectomy (N=35) | LSC Hysterectomy (N=35)
Blood transfusion (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 9 (9)

LIMITATIONS AND CAVEATS:
Data on sexual well-being will be analysed at a later date.

We received the 6 month study questionnaire of the last recruited participant A53 on 15-07-2017. We noted this date as the actual study completion date in the trial register. Although the secondary outcomes at 6 months of this last patient were received one month earlier due to the very timely sending of the questionnaire by our study secretary we decided to consider them as valid, since only secondary outcomes were collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-12-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT02631837/Prot_001.pdf
  • Statistical Analysis Plan (2016-01-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT02631837/SAP_000.pdf